CLINICAL TRIAL: NCT01562912
Title: The Prospective, Multicenter Canadian Atrial Fibrillation PVAC Cohort Study
Brief Title: Efficiency Study Evaluating the Use of PVAC Catheter Technology for Performing Ablation in Pts With Atrial Fibrillation
Acronym: CAPCOST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newmarket Electrophysiology Research Group Inc (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NERG-01
Record Dates: First submitted 2012-02-20; First posted 2012-03-26 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Atrial Fibrillation
Keywords: radiofrequency; ablation; atrial fibrillation; PVAC
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): Radiofrequency Ablation Procedure. Subjects who are undergoing AF ablation with traditional ablation technology at the same centers by the same operators. Control patients will be enrolled in a 1:2 ratio compared to the PVAC cohort. Intervention is the use of Radiofrequency Ablation.
  Interventions: Device: Radiofrequency Ablation Procedure
- PVAC Ablation Procedure (Experimental): Intervention is the use of PVAC technology. The PVAC is deployed in the left atrium over a 0.032-inch guidewire inside the PV and advanced until it is wedged within the antrum proximal to the ostium. Energy is delivered through selected electrode pairs with local potentials as well as adjacent electrode pairs, allowing bipolar current to flow to the target electrode(s) from both sides. Each application lasts for 60 seconds. When the temperature does not rise above 50°C within 15 seconds, the application should be discontinued to improve position. The PVAC may be manipulated within the antrum to ablate in a pattern of overlapping circular lesions.
  Interventions: Device: PVAC Ablation Procedure

INTERVENTIONS:
Device: Radiofrequency Ablation Procedure — Application of radiofrequency energy will be delivered during PV antral isolation procedure and should be performed with a standard, open irrigated ablation catheter and a mapping system as the investigator would perform the procedure normally.
  Other Names: THERMOCOOL Catheter, Biosense Webster; EnSite NavX Velocity, St Jude; LASSO Circular Mapping Catheter, Biosense Webster
  Arms: Control
Device: PVAC Ablation Procedure — Application of radiofrequency energy with the Pulmonary Vein Ablation Catheter(PVAC)to eliminate potentials arising from the pulmonary veins.
  Other Names: PVAC Catheter, Medtronic Inc., Ablation Frontiers
  Arms: PVAC Ablation Procedure

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia affecting the Canadian population. AF is associated with increased risk of stroke,HF, and even mortality. AF can cause debilitating symptoms, adversely affect patient's (pt's) quality of life and functional status. Hence a strategy of sinus rhythm (SR) may be pursued over a strategy of allowing AF to persist. Percutaneous catheter ablation is an effective alternative to antiarrhythmic drugs (AAD) for maintaining SR. The success rate of PV isolation off AAD is about 80-90% in pt's with PAF, but repeat procedures are required in up to 40% of pt's. After one ablation, the success rate may only be 50-70% off drugs.Current standard ablation procedures for PV antral isolation employ mapping systems which reconstructions of the LA and PV anatomy are created. Visualization may be supplemented by integration of CT/ MRI images and/or intracardiac echocardiography. Robotic navigation has been employed to assist in ablation. Based on single point unipolar radiofrequency (RF) ablation catheter where lesions are created point-by-point around the PVs to obtain electrical isolation.This results in lengthy complex, costly procedures,often more than 4 hours, which requires high degree of operator skill.Creation of contiguous, transmural lesions is challenging with standard single-point RF. A novel multipolar catheter ablation system has been evaluated for achieving PV isolation (PVAC catheter, Medtronic Inc.) An over-the-wire circular mapping/ablation catheter can be advanced into the PV antrum, and multiple lesions around the circumference of the catheter can be delivered simultaneously using duty-cycled unipolar and bipolar RF energy. Early reports, the system can achieve complete PV isolation with reduced fluoroscopy and procedural times using lower powers to achieve more reliable lesion sets.Long-term efficacy also seems comparable to standard RF ablation.This novel technology has potential to broaden the application of AF ablation, making procedures less time-consuming, less complex without compromising procedural efficacy. Published data PVAC technology outcomes are limited to studies with small sample sizes of 12-102 pt's. Data has been restricted to a small number of European centers performing moderate numbers of PVAC procedures. There is no prospective, multicenter data. Little is known about the efficiency of PVAC procedures, allowing for an assessment of cost-effectiveness in using this technology.

DETAILED DESCRIPTION:
This is a multicenter, open label, prospective, cohort study. Patients undergoing ablation with PVAC technology in up to 15 centers across Canada will be enrolled, ablated, and followed for one year post-ablation. Both primary and secondary objectives of the study will be determined from this cohort of patients. Comparisons to the traditional ablation methods will be made by collecting data from a prospective group of control subjects who are undergoing AF ablation with traditional ablation technology at the same centers by the same operators. Control patients will be enrolled in a 1:2 ratio compared to the PVAC cohort. While the final ratio of control to PVAC patients must be 1:2 by study end for each operator, the ratio may vary while the study is conducted to allow some flexibility in patient recruitment. However, the absolute difference between [# of PVAC patients] and 2x[# control patients] should not exceed 5 at any given time for any operator in any study center

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or greater.
* Patients undergoing first-time catheter ablation for AF.
* Patients with paroxysmal AF. Paroxysmal AF will be defined as self-terminating episodes less than 7 days duration. Patients should have had at least 3 episodes of AF in a one year period.
* Patients with symptomatic AF that is refractory to at least one antiarrhythmic medication. "Symptomatic" patients are those who have been aware of their AF anytime within the last 5 years prior to enrollment. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, or any combination of the above.
* At least one episode of AF must have been documented by ECG, Holter, loop recorder, telemetry, or transtelephonic monitoring within 24 months of enrollment in the study.
* Patients must be able and willing to provide written informed consent to participate in the clinical study.

Exclusion Criteria:

* Patients with persistent AF (defined as an episode of AF lasting >7 days).
* Patients with AF felt to be secondary to an obvious reversible cause.
* Patients with contraindications to systemic anticoagulation with heparin or warfarin or a direct thrombin inhibitor.
* Patients who have previously undergone AF ablation.
* Patients with left atrial size >/= 55 mm (2D echocardiography, parasternal long axis view).
* Patients who are or may potentially be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2012-02; Primary Completion 2017-12 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Procedure Duration and Fluoroscopy time | At the time of the initial ablation procedure and repeat ablations.
  Length of procedure measure in hours/minutes and use of fluoroscopy measured in minutes

SECONDARY OUTCOMES:
Incidence of emergency room visits, hospitalizations and urgent clinic visits. | 1 year follow-up post ablation
  Incidence of emergency room visits, hospitalizations and urgent clinic visits one year prior to ablation and 3, 6, 9, and 12 months post ablation.
Quality of Life measurements (CCS-SAF, AFEQT and SF-12) | 1 year post ablation
  Quality of Life measurements (CCS-SAF , AFEQT and SF-12) questionnaires at baseline, 3, 6 , 9 and 12 months.
Total ablation procedure costs. | 1 year post ablation
  calculation of procedural costs

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — Newmarket Electrophysiology Research Group
Locations (6):
- Canada (6):
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Center, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Hôpital Sacré-Coeur de Montréal, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: Undecided
to be determined

REFERENCES:
- [Derived] Essebag V, Azizi Z, Alipour P, Khaykin Y, Leong-Sit P, Sarrazin JF, Sturmer M, Morillo C, Terricabras M, Amit G, Roux JF, Patterson S, Verma A. Relationship between quality of life and burden of recurrent atrial fibrillation following ablation: CAPCOST multicentre cohort study. Europace. 2020 Jul 1;22(7):1017-1025. doi: 10.1093/europace/euaa066. PMID 32531030